CLINICAL TRIAL: NCT00900796
Title: Success and Failure of Biological Therapy: Predictors of Response in Patients With Active Ankylosing Spondylitis
Brief Title: Study Evaluating Predictors of Response in Patients With Ankylosing Spondylitis
Acronym: PRETEA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A3-4452; B1801100
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-05

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis;predictive factors
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Treatment Switching

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients diagnosed with active AS who start anti-TNF therapy according to standard clinical practice.
  Interventions: Other: Treatment switching

INTERVENTIONS:
Other: Treatment switching — If the patients do not response to first AntiTNF treatment, Investigator can switch to another anti TNF.Spanish Guidelines will be provided to the investigators, which recommend stopping biologics if there is an inadequate response after 16w of therapy and switch to another biologic. Responsive patients to the first anti-TNF who continue with this first anti-TNF adjusting dose treatment according to the Spanish guidelines or investigator criteria. The doses for each Anti TNF will be done following specific SmPc and under Investiagtor criteria

SUMMARY:
The objective of this observational study is to determine the incidence of response in patients with predictive factors of major clinical response in active ankylosing spondylitis (AS) in patients who start anti-tumor necrosis factor (anti-TNF) therapy and correlate these findings in patients who switch from one to another anti-TNF due to inefficacy under usual clinical practice conditions in Spain.

DETAILED DESCRIPTION:
A sample size of 240 patients, 120 of them exposed and 120 not exposed to factors of response. Sample will be obtain from all the consecutive patients attending the rheumatology settings included in the study who fulfill the inclusion criteria

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed of active AS who will start anti-TNF therapy following standard clinical practice as per summary of product characteristics doses.
* >18 years, both genders, any disease duration
* Signature of informed consent

Exclusion Criteria:

* Previous treatment with biological therapies
* Active tuberculosis infection (local guidelines for appropriate screening and treatment of tuberculosis in the setting of anti-TNF therapy must be followed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active ankylosing spondylitis treated in rheumatology units
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Madrid, Madrid, Spain

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A3-4452&StudyName=Study%20evaluating%20predictors%20of%20response%20in%20patients%20with%20ankylosing%20spondylitis

RESULTS

PARTICIPANT FLOW:
Groups:
- Anti-tumor Necrosis Factor Agents: Participants with active ankylosing spondylitis (AS) who were prescribed with an anti-tumor necrosis factor (anti-TNF) agent, either etanercept 50 milligram (mg) once weekly or 25 mg twice weekly subcutaneously (s.c.) or infliximab infusion 5 mg per kilogram (mg/kg) body weight intravenously (IV) at Week 0, 2, 6, 14 and 22 or adalimumab 40 mg s.c. every other week in Phase 1 of the study and if no response was observed, treatment was changed as per investigator's discretion in Phase 2 of the study.
Period: Phase 1
Arm/Group | Anti-tumor Necrosis Factor Agents
Started | 132
Completed | 121
Not Completed | 11
Not completed — Lacked sufficient information | 4
Not completed — Missing information at Week 16 | 7
Period: Between Phase 1 and Phase 2
Arm/Group | Anti-tumor Necrosis Factor Agents
Started | 121
Completed | 11
Not Completed | 110
Not completed — Responded to therapy- ineligible for Ph2 | 110
Period: Phase 2
Arm/Group | Anti-tumor Necrosis Factor Agents
Started | 11
Completed | 6
Not Completed | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Groups:
- Anti-tumor Necrosis Factor Agents (Evaluable Population): Participants with active ankylosing spondylitis (AS) who were prescribed with an anti-TNF agent, either etanercept 50 milligram (mg) once weekly or 25 mg twice weekly subcutaneously (s.c.) or infliximab infusion 5 mg per kilogram (mg/kg) body weight intravenously (IV) at Week 0, 2, 6, 14 and 22 or adalimumab 40 mg s.c. every other week, in Phase 1 of the study and who were eligible for the analysis.
Arm/Group | Anti-tumor Necrosis Factor Agents (Evaluable Population)
Number analyzed (Participants) | 121
Age Continuous [Mean (Standard Deviation); unit: years] | 42.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 85

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Clinical Response
Description: Assessment of clinical response was as per investigator's discretion. Investigators were provided with the final consensus document of the Spanish Society for Rheumatology (SER) for the biological treatment of spondyloarthropathies as a guide for defining active AS, the indication of treatment with biological therapy and the assessment of response to it.
Time Frame: Week 16
Population: Analysis population included all participants enrolled in the study who gave their consent, satisfied all evaluation criteria and had information available at Week 16 after starting the first anti-TNF treatment (Phase 1).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Anti-tumor Necrosis Factor Agents (Phase 1): Participants with active ankylosing spondylitis (AS) who were prescribed with an anti-tumor necrosis factor (anti-TNF) agent, either etanercept 50 milligram (mg) once weekly or 25 mg twice weekly subcutaneously (s.c.) or infliximab infusion 5 mg per kilogram (mg/kg) body weight intravenously (IV) at Week 0, 2, 6, 14 and 22 or adalimumab 40 mg s.c. every other week in Phase 1 of the study.
Arm/Group | Anti-tumor Necrosis Factor Agents (Phase 1)
Number analyzed (Participants) | 121
percentage of participants
  Adequate Response | 90.9 [85.79 to 96.03]
  Inadequate response | 9.1 [3.97 to 14.21]

2. Secondary Outcome: Percentage of Participants With High Probability of Response and no Response Who Received Second Anti-TNF Treatment
Description: High probability of response=participants who met at least 3 of 5 criteria at start of treatment:C-reactive Protein (CRP) >15 mg/Liter (mg/L);time from onset of disease <10 years;total spinal pain >30 millimeter (mm), mean score on 100 mm visual numeric scale (VNS) for nocturnal, total spinal pain;Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) >4 centimeter (cm), mean score on 10 cm VNS for discomfort, pain, fatigue;Bath Ankylosing Spondylitis Functional index (BASFI) <4.5 cm, mean score on 10 cm VNS evaluating functional capacity. Assessment of response was per investigator.
Time Frame: Week 32
Population: Analysis population included all participants with an inadequate response, 16 weeks after starting the first anti-TNF treatment as determined by the investigator and who received second anti-TNF treatment for at least 16 weeks (Phase 2).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Anti-tumor Necrosis Factor Agents (Phase 2): Participants with active AS who did not respond to anti-TNF treatment in Phase 1 of the study, either etanercept 50 mg once weekly or 25 mg twice weekly s.c. or infliximab infusion 5 mg/kg body weight IV at Week 0, 2, 6, 14 and 22 or adalimumab 40 mg s.c. every other week, and switched to another anti-TNF treatment in Phase 2 as per investigator's discretion.
Arm/Group | Anti-tumor Necrosis Factor Agents (Phase 2)
Number analyzed (Participants) | 6
percentage of participants | 66.7 [28.95 to 104.39]

3. Secondary Outcome: Percentage of Participants With Low Probability of Response and no Response Who Received Second Anti-TNF Treatment
Description: Low probability of response = participants who met no more than 2 of 5 criteria at time of treatment start: CRP > 15 mg/L; time from onset of disease less than < 10 years; total spinal pain > 30 mm, measured as mean score on 100 mm VNS (higher score=more severe pain) for nocturnal and total spinal pain; BASDAI > 4 cm, measured as mean score on 10 cm VNS (higher score=more severe state) for discomfort, pain and fatigue; BASFI < 4.5 cm; measured as mean score on 10 cm VNS (higher score=less functionality) evaluating functional capacity. Assessment of response was as per investigator's criteria.
Time Frame: Week 32
Population: Data was not analyzed as no participant met the criteria for low probability of response in phase 2 of the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anti-tumor Necrosis Factor Agents (Phase 2)
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Participants With Low Probability of Response and a Clinical Response at Week 16
Description: as for outcome 3
Time Frame: Week 16
Population: Analysis population included all participants enrolled in study who gave their consent, satisfied all evaluation criteria and had information available at Week 16 after starting first anti-TNF treatment (Phase 1). N (number of participants analyzed) signifies those participants who had low probability of response and were evaluable for the measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anti-tumor Necrosis Factor Agents (Phase 1)
Number analyzed (Participants) | 28
percentage of participants | 96.4 [89.55 to 103.30]

5. Secondary Outcome: Percentage of Participants With Assessment in Ankylosing Spondylitis (ASAS) 40 Response at Week 16
Description: ASAS measures symptomatic improvement in ankylosing spondylitis (AS) participants ASAS = 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 40 = 40 percent (%) improvement from baseline and an absolute change of greater than or equal to (>=) 2 units on a 0-10 scale (0=no disease activity, 10=high disease activity) for >= 3 domains, and no worsening in remaining domain.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anti-tumor Necrosis Factor Agents (Phase 1)
Number analyzed (Participants) | 121
percentage of participants | 33.1 [24.68 to 41.44]

6. Secondary Outcome: Percentage of Participants Who Switched to Another Anti-TNF Treatment Due to Lack of Efficacy
Time Frame: Week 16
Population: Analysis population included all participants enrolled in the study who gave their consent, satisfied all evaluation criteria and had information available at Week 16 after starting the first anti-TNF treatment (Phase 1). Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anti-tumor Necrosis Factor Agents (Phase 1)
Number analyzed (Participants) | 11
percentage of participants | 72.7 [46.41 to 99.05]

7. Secondary Outcome: Percentage of Participants With ASAS 40 Response Who Started Second Anti-TNF Treatment and Were Treated for at Least 16 Weeks
Description: ASAS measures symptomatic improvement in ankylosing spondylitis (AS) participants ASAS = 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 40 = 40% improvement from baseline and an absolute change of greater than or equal to (>=) 2 units on a 0-10 scale (0=no disease activity, 10=high disease activity) for >= 3 domains, and no worsening in remaining domain.
Time Frame: Week 32
Population: Analysis population included all participants with an inadequate response, 16 weeks after starting the first anti-TNF treatment as determined by ASAS 40 and who received second anti-TNF treatment for at least 16 weeks (Phase 2).
Measure: Number; unit: percentage of participants
Arm/Group | Anti-tumor Necrosis Factor Agents (Phase 2)
Number analyzed (Participants) | 6
percentage of participants | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Anti-tumor Necrosis Factor Agents: Participants with active AS who were prescribed with an anti-TNF agent, either etanercept 50 mg once weekly or 25 mg twice weekly s.c. or infliximab infusion 5 mg/kg body weight IV at Week 0, 2, 6, 14 and 22 or adalimumab 40 mg s.c. every other week in Phase 1 of the study and if no response was observed, treatment was changed as per investigator's discretion in Phase 2 of the study.
Arm/Group | Anti-tumor Necrosis Factor Agents
Serious Adverse Events (participants affected / at risk) | 1/132
Other Adverse Events (participants affected / at risk) | 9/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-tumor Necrosis Factor Agents (N=132)
Tonsillar neoplasm (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-tumor Necrosis Factor Agents (N=132)
Upper respiratory tract infection (General disorders) | 3
Injection site reaction (General disorders) | 4
Gastroenteritis viral (General disorders) | 1
Diarrhoea and vomiting (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.